CLINICAL TRIAL: NCT03775434
Title: An Open-label, Multicenter, Phase Ib Study of B244 Delivered as a Topical Spray to Assess Safety in Pediatric Subjects Aged 2 to 17 Years With Atopic Dermatitis
Brief Title: A Study of B244 Delivered as a Topical Spray to Assess Safety in Pediatric Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADB244-002
Record Dates: First submitted 2018-12-07; First posted 2018-12-14 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Eczema; Atopic Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: All subjects will receive active product
Masking Description: This is a single arm open label study. Subjects will be assigned to the study treatment arm. Each participant will be scheduled to receive investigational product (IP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B244 (Experimental): B244 suspension in 30ml/bottle
  Interventions: Drug: Experimental: B244

INTERVENTIONS:
Drug: Experimental: B244 — B244 suspension in 30ml/bottle

SUMMARY:
An open-label, multicenter, Phase Ib study of B244 delivered as a topical spray to assess safety in pediatric subjects aged 2 to 17 years with atopic dermatitis

Condition or disease Intervention/treatment Phase Atopic Dermatitis (Eczema) Biological: B244 Phase 1b

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, single arm, multiple site study assessing twice daily B244 application for 28 days in pediatric subjects with mild to moderate atopic dermatitis.

Number of Subjects:

The study will enroll 36 subjects in 3 cohorts of 12 subjects:

* Cohort 1: subjects aged 2 to 5 years.
* Cohort 2: subjects aged 6 to 11 years.
* Cohort 3, subjects aged 12 to 17 years.

At Screening and Baseline, all subjects must have confirmed diagnosis of atopic dermatitis, as defined by the Hanifin and Rajka criteria, which involves a minimum of 10% but no more than 60% body surface area and a Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) scale of 2 or 3.

The duration of the study will be approximately 7 weeks. Subjects will attend for a Screening visit between Days -21 and -14. If all eligibility criteria and none of the exclusion criteria are met, subjects will be enrolled into the study and will be required to undergo a 14 day washout period (Days-14 to -1). Subjects will attend the study center on Day 1 and the Baseline assessments will be performed before application of the first dose.

On confirmation of continued eligibility the subject and parent or guardian of the subject will be coached on how to apply medication, depending on the affected areas. They will be instructed to apply B244 twice daily (approximately 12 hours apart) for 28 days.

The first dose will be applied in the clinic under the supervision of clinical staff. Details of dose administration will be recorded in the study diary provided. The subjects with their parent or guardian will return to the study center on Days 7, 14, and 21 for completion of study assessments.

There will be a final study visit on Day 28, this will be defined as the end of the study for the subjects. A time window of ±2 day will be permitted for these 4 visits. There will not be a period of confinement in the study center all visits will be outpatient visits. Safety monitoring will include review of TEAEs, vital signs and physical examination. Efficacy will be assessed using EASI, vIGA-AD scale, POEM and ItchMan scores.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to be included in the study only if all of the following criteria apply:

  1. Male and female subjects 2 to 17 years of age, inclusive.
  2. Confirmed diagnosis of atopic dermatitis according to the Hanifin and Rajka criteria.
  3. A minimum of 10% but no more than 60% of the subjects' body surface area (see Appendix 6 for guidance) is affected by atopic dermatitis (affected is defined by physical examination findings: erythema, edema, scaling, lichenification, and excoriation; with the excoriation serving as the physical examination correlate of pruritus).
  4. A vIGA-AD scale of 2 or 3 at Screening and Baseline.
  5. Subject, or the parent or guardian, to provide written informed consent and authorization for protected health information disclosure.
  6. Subjects must be generally in good health based on Investigator's assessment (other than atopic dermatitis).
  7. Normal vital signs, or with no clinically significant vital signs that in the opinion of the Investigator, would place the subject at increased risk or would confound the objectives of the study.
  8. Females must not be pregnant, as confirmed by negative urine pregnancy testing. Female subjects aged ≥11 years old, or female patients <11 years old who have started menstruating, will have urinary pregnancy test performed at Screening and prior to the first dose with negative results in order to participate in the study. Females must either practice abstinence from heterosexual contact or use one of the highly effective contraceptive options described in the Appendix 5.
  9. Male subjects of reproductive potential, must be willing to practice effective contraception during the study while receiving study treatment from Day 1 and for 7 days after the last study visit (Day 28).
  10. Ability to comprehend and comply with study procedures.
  11. Agree to commit to participate in the current protocol.
  12. Provide written informed consent prior to any study procedure being performed.

      Exclusion Criteria:

      Subjects are excluded from the study if any of the following criteria apply:

  <!-- -->

  1. Clinically significant physical or mental disorder which, in the opinion of the Investigator, would place the subject at increased risk or would confound the objectives of the study.
  2. Subjects with atopic dermatitis on the face only.
  3. Active cutaneous bacterial, viral or fungal infection in any treatment area at Baseline (eg, clinically infected atopic dermatitis).
  4. History or presence of immunological deficiencies or diseases, organ transplant, human immunodeficiency virus (HIV), diabetes, malignancy, malignant or pre-malignant skin conditions, serious active or recurrent infection, systemic immunosuppressive regimens, clinically significant renal disease severe hepatic disorders, or other severe uncontrolled conditions (eg, drug or alcohol abuse), that are significant and/or that may pose a health risk to the subject in the study or may have an impact on the study assessments.
  5. Unstable atopic dermatitis or a consistent requirement for high-potency corticosteroids (class I-III steroids).
  6. Active systemic or localized infection (including infected AD).
  7. Subjects unable to comply with the excluded medication/therapy restriction
  8. Known hypersensitivity to the study treatment.
  9. Known to have hepatitis B, hepatitis C or HIV I or II tests. Details will be recorded in medical history, a blood sample will not be collected for confirmation.
  10. Female subject who is pregnant, breastfeeding, or considering pregnancy during the study.
  11. Any skin condition which in the Investigator's opinion may interfere with the evaluation of atopic dermatitis.
  12. Use of any investigational drugs within the previous 30 days prior to dosing or within a period of less than 5 times the drug's half-life, whichever is longer.
  13. Use of any biologic within a period of 5 times its half-life.
  14. Children or relatives of the Sponsor, clinical research organization, or the Study Site personnel are excluded from participating in the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ng-Cashin, MD, Study Director — Chief Medical Officer; Spiros Jamas, ScD, Study Director — AOBiome Therapeutics
Locations (6):
- United States (6):
  - Dermatology Trial Associates, Bryant, Arkansas
  - L.A. Universal Research Center, Inc., Los Angeles, California
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Virginia Clinical Research, INC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B244: B244 suspension in 30ml/bottle.
  B244: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
Period: Overall Study
Arm/Group | B244
Started | 28
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: ITT population: All subjects who were enrolled and took at least 1 dose of study treatment.
Arm/Group | B244
Number analyzed (Participants) | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 7.4 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Percentage of Total Body Surface Area Affected by Atopic Dermatitis [Mean (Standard Deviation); unit: % of total body surface area] — Body Surface Area (BSA) ranges from 0% to 100% with higher values representing a greater extent of atopic dermatitis. Affected area is defined by physical examination findings: erythema, edema, scaling, lichenification, and excoriation; with the excoriation serving as the physical examination correlate of pruritus.
  % of total body surface area | 17.98 (7.581)
Baseline vIGA-AD Score [Count of Participants; unit: Participants] — The vIGA-AD is a physician assessment ranking of Atopic Dermatitis symptoms from 0-clear, to 4- severe.
  Participants
    2=Mild | 11
    3=Moderate | 17
Weight [Mean (Standard Deviation); unit: kg] | 36.22 (30.599)
Height [Mean (Standard Deviation); unit: cm] | 124.0 (29.95)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.5 (7.73)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all adverse events reporting from Baseline to Day 28.
Time Frame: Baseline to Day 28
Population: ITT population: All subjects who were enrolled and took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | B244
Number analyzed (Participants) | 28
Participants | 11

2. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Exam.
Description: A physical exam will be conducted by a physician assessing systems (General appearance, Dermatological, Musculoskeletal, Thyroid, HEENT [Head, eyes, ears, nose, throat], Lymphatic, Respiratory, Gastrointestinal, Cardiovascular, Neurological, Extremities, and other). Clinical significance of the physical exam will be determined at investigator's discretion. Results for each system were assessed as Normal, Abnormal CS (clinically significant), or Abnormal NCS (not clinically significant) and shift was analyzed from Baseline to Day 28.
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all subjects who were enrolled and took at least 1 dose of study treatment) that remained in the study at Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | B244
Number analyzed (Participants) | 25
Participants
  Cardiovascular: Normal -> Normal | 25
  Dermatological: Normal -> Abnormal CS | 1
  Dermatological: Normal -> Normal | 24
  Extremities: Normal -> Normal | 25
  Gastrointestinal: Normal -> Normal | 25
  General Appearance: Abnormal NCS -> Abnormal NCS | 1
  General Appearance: Normal -> Normal | 24
  HEENT: Abnormal CS-> Normal | 1
  HEENT: Normal -> Normal | 24
  Lymphatic: Normal -> Normal | 25
  Musculoskeletal: Normal -> Normal | 25
  Neurological: Normal -> Normal | 25
  Respiratory: Normal -> Abnormal NCS | 1
  Respiratory: Normal -> Normal | 24
  Thyroid: Missing -> Normal | 1
  Thyroid: Normal -> Normal | 24

3. Primary Outcome: Mean Change in Blood Pressure From Baseline at Day 28
Description: Blood pressure will be obtained (mmHg). Clinical significance of blood pressure will be determined at the investigator's discretion. Change from Day 28 to Baseline.
Time Frame: Baseline to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | B244
Number analyzed (Participants) | 25
mmHg
  Diastolic Blood Pressure | 1.6 (9.3)
  Systolic Blood Pressure | 1.8 (10.8)

4. Other Pre Specified Outcome: Changes in the Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD).
Description: The vIGA-AD is a physician assessment ranking of Atopic Dermatitis symptoms from 0-clear, to 4- severe.
Time Frame: Baseline, Days 7, 14, 21, and 28
Population: Subjects from the Intent to Treat (ITT) population (all subjects who were enrolled and took at least 1 dose of study treatment) that remained in the study at each respective visit day.
Measure: Count of Participants; unit: Participants
Arm/Group | B244
Number analyzed (Participants) | 28
Participants
  Change from Baseline on Day 7: number analyzed (Participants) | 26
  Change from Baseline on Day 7: 4 - Worsen by 4 grades | 0
  Change from Baseline on Day 7: 3 - Worsen by 3 grades | 0
  Change from Baseline on Day 7: 2 - Worsen by 2 grades | 0
  Change from Baseline on Day 7: 1 - Worsen by 1 grade | 2
  Change from Baseline on Day 7: No change | 23
  Change from Baseline on Day 7: -1 - Improved by 1 grade | 1
  Change from Baseline on Day 7: -2 - Improved by 2 grades | 0
  Change from Baseline on Day 7: -3 - Improved by 3 grades | 0
  Change from Baseline on Day 7: -4 - Improved by 4 grades | 0
  Change from Baseline on Day 14: number analyzed (Participants) | 25
  Change from Baseline on Day 14: 4 - Worsen by 4 grades | 0
  Change from Baseline on Day 14: 3 - Worsen by 3 grades | 0
  Change from Baseline on Day 14: 2 - Worsen by 2 grades | 0
  Change from Baseline on Day 14: 1 - Worsen by 1 grade | 2
  Change from Baseline on Day 14: No change | 20
  Change from Baseline on Day 14: -1 - Improved by 1 grade | 3
  Change from Baseline on Day 14: -2 - Improved by 2 grades | 0
  Change from Baseline on Day 14: -3 - Improved by 3 grades | 0
  Change from Baseline on Day 14: -4 - Improved by 4 grades | 0
  Change from Baseline on Day 21: number analyzed (Participants) | 25
  Change from Baseline on Day 21: 4 - Worsen by 4 grades | 0
  Change from Baseline on Day 21: 3 - Worsen by 3 grades | 0
  Change from Baseline on Day 21: 2 - Worsen by 2 grades | 0
  Change from Baseline on Day 21: 1 - Worsen by 1 grade | 2
  Change from Baseline on Day 21: No change | 17
  Change from Baseline on Day 21: -1 - Improved by 1 grade | 6
  Change from Baseline on Day 21: -2 - Improved by 2 grades | 0
  Change from Baseline on Day 21: -3 - Improved by 3 grades | 0
  Change from Baseline on Day 21: -4 - Improved by 4 grades | 0
  Change from Baseline on Day 28: number analyzed (Participants) | 25
  Change from Baseline on Day 28: 4 - Worsen by 4 grades | 0
  Change from Baseline on Day 28: 3 - Worsen by 3 grades | 0
  Change from Baseline on Day 28: 2 - Worsen by 2 grades | 0
  Change from Baseline on Day 28: 1 - Worsen by 1 grade | 2
  Change from Baseline on Day 28: No change | 17
  Change from Baseline on Day 28: -1 - Improved by 1 grade | 5
  Change from Baseline on Day 28: -2 - Improved by 2 grades | 1
  Change from Baseline on Day 28: -3 - Improved by 3 grades | 0
  Change from Baseline on Day 28: -4 - Improved by 4 grades | 0

5. Other Pre Specified Outcome: Changes in Area Severity Index (EASI) Score.
Description: EASI is a validated tool used to measure the severity and extent of atopic dermatitis where clinical investigators assess the presence and severity of erythema, edema/papulation, excoriation, and lichenification (score 0-3: none=0, mild=1, moderate=2, severe=3, half-points allowed) and area of involvement (score 0-6: 0=0% involvement, 1=1-9% involvement, 2=10-29% involvement, 3=30-49% involvement, 4=50-69% involvement, 5=70-89% involvement, 6=90-100% involvement) across head and neck, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks). The EASI score can range from 0.0 to 72.0 with increments of 0.1 and higher scores representing a greater severity of atopic dermatitis.
Time Frame: Baseline, Days 7, 14, 21, and 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244
Number analyzed (Participants) | 28
score on a scale
  Change from Baseline to Day 7: number analyzed (Participants) | 26
  Change from Baseline to Day 7 | -0.31 (2.920)
  Change from Baseline to Day 14: number analyzed (Participants) | 25
  Change from Baseline to Day 14 | -1.30 (4.088)
  Change from Baseline to Day 21: number analyzed (Participants) | 25
  Change from Baseline to Day 21 | -1.98 (4.693)
  Change from Baseline to Day 28: number analyzed (Participants) | 25
  Change from Baseline to Day 28 | -2.31 (4.109)

6. Other Pre Specified Outcome: Changes in Patient Oriented Eczema Measure (POEM Total Score).
Description: POEM is a survey that consists of 7 questions that assesses the quality of life of patient's with eczema to determine their disease severity. The 7 questions are scored out of 4 points based on frequency of occurrence during the prior week (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days). A higher total score indicates a higher severity of disease (0 [clear] to 28 [very severe]).
Time Frame: Baseline, Days 7, 14, 21, and 28
Population: ITT population: All subjects who were enrolled and took at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244
Number analyzed (Participants) | 28
score on a scale
  Change from Baseline to Day 7: number analyzed (Participants) | 26
  Change from Baseline to Day 7 | -1.2 (4.68)
  Change from Baseline to Day 14: number analyzed (Participants) | 25
  Change from Baseline to Day 14 | -4.2 (5.21)
  Change from Baseline to Day 21: number analyzed (Participants) | 25
  Change from Baseline to Day 21 | -4.4 (6.10)
  Change from Baseline to Day 28: number analyzed (Participants) | 25
  Change from Baseline to Day 28 | -4.2 (7.03)

7. Other Pre Specified Outcome: Changes in Patient Reported Outcome (Self-reported ItchMan Scale).
Description: The Burn Man Itch Scale is used as a self report tool for subjects to indicate how itchy the area of atopic dermatitis feels at the timepoints during the study. It's reported on a scale between 0-comfortable, no itch and 4-Itches most terribly; impossible to sit still; concentrate.
Time Frame: Baseline, Days 7, 14, 21, and 28
Population: ITT population: All subjects who were enrolled and took at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244
Number analyzed (Participants) | 28
score on a scale
  Change from Baseline to Day 7: number analyzed (Participants) | 26
  Change from Baseline to Day 7 | -0.2 (0.92)
  Change from Baseline to Day 14: number analyzed (Participants) | 25
  Change from Baseline to Day 14 | -0.8 (1.20)
  Change from Baseline to Day 21: number analyzed (Participants) | 25
  Change from Baseline to Day 21 | -0.6 (1.26)
  Change from Baseline to Day 28: number analyzed (Participants) | 25
  Change from Baseline to Day 28 | -0.8 (1.40)

8. Primary Outcome: Mean Change in Pulse Rate From Baseline at Day 28
Description: Pulse rate (beats per minute [bpm]) will be obtained. Clinical significance of pulse rate will be determined at the investigator's discretion. Change from Day 28 to Baseline.
Time Frame: Baseline to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | B244
Number analyzed (Participants) | 25
bpm | 3.9 (15.3)

9. Primary Outcome: Mean Change in Body Temperature From Baseline at Day 28
Description: Body temperature (°C) will be obtained. Clinical significance of body temperature will be determined at the investigator's discretion. Change from Day 28 to Baseline.
Time Frame: Baseline to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | B244
Number analyzed (Participants) | 25
°C | -0.2 (0.6)

ADVERSE EVENTS:
Time Frame: Baseline to Day 28
Description: All AEs and SAEs will be collected from Baseline until the final visit or Early Termination Visit. All SAEs will be recorded and reported to the Sponsor or designee within 24 hours. The Investigator or designee will submit any updated SAE data to the Sponsor within 24 hours of it being available.
Arm/Group | B244
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 (N=28)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Localized infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 60 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional 90 days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03775434/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03775434/SAP_001.pdf